CLINICAL TRIAL: NCT03521453
Title: PEPPER : PErcePtion of Pre-anesthesia Visit With or Without Robot
Acronym: PEPPER
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PEPPER-01
Record Dates: First submitted 2018-03-01; First posted 2018-05-11 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Satisfaction, Personal; Anesthesia
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: Conventionnel written information
- After, with PEPPER: Written information + presence of a robot (PEPPER) in the waiting room, who will give informations.
  Interventions: Other: PEPPER robot

INTERVENTIONS:
Other: PEPPER robot — Presence of a Robot (PEPPER Robot), designed and programmed to give informations, using a screen and vocal. All the patients in the second period will have access to,the robot, while waiting for the visit.
  Groups: After, with PEPPER

SUMMARY:
Pre-anesthesia visit for scheduled surgery is mandatory by law in France. During this visit, patients should be informed of the different available technics of anesthesia (i.e. general or loco-regional) and of their own risks .

Nowadays, many informations are given through written paper and leaflets, just before the consultation. In addition, patients need usually to wait for the doctor. This time may be used to give information, and new information's support, such as videos, may be used.

The aim of this study is to evaluated if a robot (PEPPER), who is able to answer to patients and to give informations, may increase the satisfaction of patients having a pre anesthesia visit for a scheduled surgery.

DETAILED DESCRIPTION:
Before- after observational study.

All adult patients (age≥18 yrs) coming for a pre-anesthesia visit will be proposed to fulfill a questionnaire regarding their satisfaction and the quality of information they received.

* in the first period, patients will receive paper informations before the anesthesia visit.
* in the second period, they will have the same paper informations but a robot PEPPER will also stand in the waiting room and propose to the patients to give them informations about anesthesia, patients journey, risks, blood transfusion etc...

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for a pre-Anesthesia visit during the study period

Exclusion Criteria:

* Refusal to answer the questionnaire
* unable to answer the questionnaire (not speaking french...)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients scheduled for a pre-Anesthesia visit during the study period (for orthopedic, general, urologic, ophthalmologic surgeries or for endoscopic examination under anesthesia).
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Patients satisfaction about the pre-anesthesia visit | 1 hour
  numerical scale from 0 to 10 (poor to excellent)

SECONDARY OUTCOMES:
quality of information | 1 hour
  numerical scale from 0 to 10 (poor to excellent)
quality of information about risks | 1 hour
  numerical scale from 0 to 10 (poor to excellent)
annoying of waiting | 1 hour
  numerical scale from 0 to 10 (none to maximal)

CONTACTS AND LOCATIONS:
Overall Officials: sigismond Lasocki, MD, PhD, Study Chair — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No